CLINICAL TRIAL: NCT03986762
Title: A Phase IA Open Label Pharmaco- Magnetic Resonance Spectrography (MRS) Study of Clavulanic Acid Daily Repeated Administration in Remitted Cocaine Use Disorder Subjects
Brief Title: Open Label Pharmaco- Magnetic Resonance Spectrography (MRS) Study of Clavulanic Acid
Acronym: CLAVMRPilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25506
Record Dates: First submitted 2019-02-15; First posted 2019-06-14 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Cocaine Dependence, in Remission; Cocaine Abuse, in Remission; Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Clav (Experimental)
  Interventions: Drug: Clavulanic Acid

INTERVENTIONS:
Drug: Clavulanic Acid — ~10 days of Clavulanic Acid

SUMMARY:
The main purpose of this study is to determine how the study drug, clavulanic acid, affects glutamate in the brain using Magnetic Resonance (MR/MRI) scans. In this study, subjects will receive the study drug, clavulanic acid and undergo 4 MRI scans. This is being studied to determine the correct dosing of clavulanic acid, and to gather data so future studies can be done to find out if this drug is helpful in treating cocaine dependence. Currently, there is no available medication treatment for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for cocaine use disorder, moderate to severe in early remission.
* Be male or female adult volunteers ages 18-65 inclusive.
* If female and of childbearing potential, must have a negative pregnancy test within 48 hours of beginning the study and be willing to use acceptable contraception or be abstinent for 14 days prior to study, through the entire study and 30 days after study participation.

Exclusion Criteria:

* Be unable to complete an MRI scan

(For full inclusion/exclusion criteria or for more information, please contact the site directly.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Glutamate change from baseline | 10-17 Days
  Change in brain glutamate concentration at Day 10-17 compared with baseline.
Glutamate/creatine ratio change from baseline | 10-17 Days
  Change in brain glutamate/creatine ratio at Day 10-17

SECONDARY OUTCOMES:
Glutamate change after dose stoppage | Day 10-11
  Change in brain glutamate concentration in 2 brain areas associated with addiction at Day 11 compared with Day 10.
Glutamate/creatine ratio change after dose stoppage | Day 10-11
  Change in brain glutamate/creatine ratio in 2 brain areas associated with addiction at Day 11 compared with Day 10.
Change in brain glutamine from baseline | 10-17 Days
  Change in brain glutamine concentration in 2 brain areas at Day 10-17 compared with baseline.
Change in brain glutamine/creatine ratio from baseline | 10-17 Days
  Change in glutamine/creatine ratio in 2 brain areas at Day 10-17 compared with baseline.
Number of participants with treatment-related adverse events (AEs) as assessed by comprehensive metabolic panel, complete blood count, ekg, urinalysis, C-SSRS, and any self-reported change in health. | 1-31 days (during and after study dosing period)
  Adverse events (AES) will be defined as any clinically significant changes in vital signs, indications of suicidal ideation or behavior on the Columbia Suicide Severity Rating Scale (C-SSRS), clinically significant change in Electrocardiogram (EKG) parameters and clinically significant changes in laboratory bloodwork (Complete blood count, comprehensive metabolic panel, urinalysis), or any self reported side effects compared with baseline.
  AEs will be collected throughout the study and reviewed by a physician. An evaluation of AE severity (mild, moderate, severe) will be evaluated by a physician based on participant self-report. AEs per subject will be listed by organ system, and the number of AEs within the subject population will be totaled.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Morrison, M.D., Principal Investigator — Temple University
Locations (1):
- Episcopal Hospital Medical Arts Building, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Uys JD, LaLumiere RT. Glutamate: the new frontier in pharmacotherapy for cocaine addiction. CNS Neurol Disord Drug Targets. 2008 Nov;7(5):482-91. doi: 10.2174/187152708786927868. PMID 19128205
- [Background] Rasmussen BA, Baron DA, Kim JK, Unterwald EM, Rawls SM. beta-Lactam antibiotic produces a sustained reduction in extracellular glutamate in the nucleus accumbens of rats. Amino Acids. 2011 Feb;40(2):761-4. doi: 10.1007/s00726-010-0589-0. Epub 2010 Apr 13. PMID 20383795
- [Background] Ward SJ, Rasmussen BA, Corley G, Henry C, Kim JK, Walker EA, Rawls SM. Beta-lactam antibiotic decreases acquisition of and motivation to respond for cocaine, but not sweet food, in C57Bl/6 mice. Behav Pharmacol. 2011 Aug;22(4):370-3. doi: 10.1097/FBP.0b013e3283473c10. PMID 21543969
- [Background] Kovalevich J, Corley G, Yen W, Rawls SM, Langford D. Cocaine-induced loss of white matter proteins in the adult mouse nucleus accumbens is attenuated by administration of a beta-lactam antibiotic during cocaine withdrawal. Am J Pathol. 2012 Dec;181(6):1921-7. doi: 10.1016/j.ajpath.2012.08.013. Epub 2012 Sep 29. PMID 23031254
- [Background] Ramadan S, Lin A, Stanwell P. Glutamate and glutamine: a review of in vivo MRS in the human brain. NMR Biomed. 2013 Dec;26(12):1630-46. doi: 10.1002/nbm.3045. Epub 2013 Oct 4. PMID 24123328